CLINICAL TRIAL: NCT00829387
Title: Cognitive Behavioral Therapy for Diabetic Peripheral Neuropathic Pain
Brief Title: Cognitive Behavioral Therapy for Diabetic Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B6044R; RK0035 (Other: VACHS)
Record Dates: First submitted 2009-01-24; First posted 2009-01-27 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Diabetic Peripheral Neuropathic Pain
Keywords: Diabetes; Pain; Neuropathic Pain
MeSH Terms: conditions — Diabetes Mellitus; Pain; Neuralgia | interventions — Cognitive Behavioral Therapy; Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral (Experimental): Cognitive behavioral therapy - Ten sessions of individual treatment delivered by a doctoral level psychologist.
  Interventions: Behavioral: CBT plus standard pharmaceutical care (CBT/SC)
- Educational (Active Comparator): Diabetes Education - Ten individual sessions of diabetes educations delivered by a doctoral level psychologist under the supervision of a certified diabetes educator
  Interventions: Behavioral: Diabetic Education plus standard pharmaceutical care (ED/SC)

INTERVENTIONS:
Behavioral: CBT plus standard pharmaceutical care (CBT/SC) — Ten sessions of individual treatment delivered by a doctoral level psychologist.
  Other Names: cognitive behavioral therapy
  Arms: Behavioral
Behavioral: Diabetic Education plus standard pharmaceutical care (ED/SC) — Ten individual sessions of diabetes educations delivered by a doctoral level psychologist under the supervision of a certified diabetes educator.
  Other Names: patient education
  Arms: Educational

SUMMARY:
The purpose of this study is to evaluate the efficacy of a brief psychological intervention, cognitive-behavior therapy, for the management of persistent pain associated with diabetic peripheral neuropathic pain.

DETAILED DESCRIPTION:
Research Design: A randomized controlled design will be employed in which CBT plus standard pharmaceutical care (CBT/SC) is compared to an educational intervention plus standard pharmaceutical care (ED/SC) treatment condition. A target sample size of approximately 215 participants will be recruited. Participants will be randomized in equal numbers to the two conditions.

Methodology: Study participants will be evaluated pre-treatment (baseline), 12 weeks post-baseline (post-treatment) and at 36 weeks post-baseline (follow-up). Baseline assessment will include a physical examination to confirm the diagnosis of diabetic neuropathy. The primary outcome measure will be pain intensity. Secondary outcome measures will be pain quality, pain-related disability, and physical and emotional functioning. Measures of treatment feasibility will also be examined. CBT and ED will be provided in 10 weekly, individual treatment sessions of 60 minutes. The effectiveness of the randomization process will be tested by examining potential between condition differences on important demographic and pain-relevant descriptive variables, as well as on the dependent measures. Analyses of covariance will be employed to determine whether statistically significant differences in the two treatment conditions are observed at the 12- and 36-week intervals controlling for pretreatment/baseline scores on these same measures and other covariates identified previously.

Hypotheses Treatment outcome hypotheses

* Persons with DPNP receiving cognitive behavioral therapy with standard pharmaceutical care (CBT/SC), relative to those receiving diabetic education with standard pharmaceutical care (ED/SC), will demonstrate, immediately following treatment improvements on several measures of the experience of persistent pain, including pain intensity, pain quality, pain-related disability, sleep quality, physical functioning, and emotional functioning, and they will have fewer added pain medication doses and concomitant pain treatments.
* Persons with DPNP receiving CBT/SC, relative to those receiving ED/SC, will demonstrate maintenance of these benefits at a 36-week post-baseline follow-up period.

Treatment satisfaction and feasibility hypotheses

- Persons with DPNP receiving CBT/SC, relative to those receiving ED/SC, will demonstrate, immediately following treatment higher ratings of treatment credibility and treatment satisfaction, and higher rates of treatment session attendance and lower rates of treatment dropout.

Exploratory secondary analyses of predictors of treatment participation and outcome

* Increased readiness to adopt a self-management approach will be positively associated with higher ratings of treatment credibility and treatment satisfaction, higher rates of treatment session attendance and lower rates of treatment dropout, and for participants in the CBT condition only, higher rates of adherence to therapist recommendations for pain coping skill practice and other intersession goals.
* Increased readiness to adopt a self-management approach over the course of treatment will be associated with improved outcomes following treatment.
* Increased readiness to adopt a self-management approach at treatment termination will significantly predict maintenance of treatment benefits on follow-up.
* Persons with medical and psychiatric comorbidities will demonstrate, relative to those without these comorbidities, less improved outcomes, lower rates of treatment session attendance and higher rates of treatment dropout, and for the CBT condition only, lower rates of adherence to therapist recommendations for pain coping skill practice and other intersession goals.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of type 2 diabetes mellitus according to American Diabetes Association criteria
* History of daily lower extremity pain or discomfort (burning, tingling or other paresthesias) for a period of at least 3 months immediately prior to enrollment,
* Presence of neuropathy, as determined by evaluation at the VACHS Neuromuscular Disease and Neuropathy Clinic at the time of the baseline examination
* Judgment of the study endocrinologist (EH) that the patient is not experiencing a paradoxical precipitation of neuropathy following institution of good control which can be expected to resolve spontaneously
* Confirmation of the study neurologists that pain is not attributable to other medical conditions that could mimic DPNP (e.g., HIV, Hepatitis C, cryoglobulinemia, pernicious anemia, untreated hypothyroidism)
* Documentation of treatment of neuropathic pain with the maximum dose of one of the medications identified as a first line or second line treatment in either VA guidelines28 or other published consensus recommendations27 with maximum dose defined as either the maximum allowable dose or the maximum tolerated dose for the recommended duration of an adequate trial, unless otherwise contraindicated or patient refusal)
* Continued use of a guideline endorsed medication for neuropathic pain (unless otherwise contraindicated or patient refusal)
* Continued refractory pain despite pharmacological intervention as described above (as determined by a pain intensity score at least 4 on a 0-10 numeric rating scale)
* No medical condition that could impair the subject's ability to participate (e.g., unstable angina, severe COPD, limb amputation, intermittent claudication)
* No psychiatric condition (e.g., active substance abuse, psychosis or suicidality) that could impair subjects' ability to participate as defined by their responses to the SCID and BDI (e.g., presence of major Depressive Disorder and BDI score 30 or greater or presence of suicidal intent; presence of these conditions will require immediate medical/psychiatric attention to assure safety and institution of appropriate treatment)
* Absence of dementia defined by a score of 24 or greater on the Folstein Mini-Mental Status Exam (MMSE)
* Urine toxicology screen confirming the absence of illegal substances or non-prescribed opioids
* Provision of participant consent to consult their primary care physician and review their medical records to ensure that eligibility criteria are met,
* Availability of a touch-tone telephone in the participant's residence to facilitate the provision of IVR data
* English fluency sufficient to participate meaningfully in treatment. Prospective participants' medical and pharmacy records will be reviewed to determine whether they meet the 4th and 5th criteria listed above.

Exclusion Criteria:

* No history of Type 2 diabetes mellitus
* Any life threatening illnesses or acute physical disease
* Any current psychiatric condition (psychosis, substance abuse/dependence)
* Any current suicidal thoughts or ideations
* The presence of profound cognitive impairment rendering successful participation in CBT or ED impossible
* prior or current psychological treatment for chronic pain
* The presence of physical disabilities resulting in an inability to attend treatment sessions and/or inability to participate in telephone interventions (e.g., severe dysarthria)
* No access to touch tone telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Kerns, PhD, Principal Investigator — VA Connecticut Healthcare System
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - VA Connecticute Health Care System, West Haven, Connecticut

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited June 2010 through March 2013 at VA Connecticut Healthcare System
Period: Overall Study
Arm/Group | Behavioral | Educational
Started | 23 | 24
Completed | 20 | 21
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Disqualified by PI | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral | Educational | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (9.12) | 60.8 (7.58) | 62.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 21 | 23 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 16 | 17 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Pain Intensity
Description: Primary outcome is the estimated mean change in pain intensity ratings from baseline to 12 weeks post-baseline comparing CBT and Educational arms
  Average pain intensity rating over the last 7 days; 0 (no pain at all) to 10 (worst pain imaginable). The higher the score, the more perceived pain a participant reported.
Time Frame: baseline to 12 weeks post-baseline [post-treatment]
Population: Not everyone that completed baseline data completed 12 week post treatment assessments; making the number of participants analyzed different than reported for baseline data only.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Behavioral | Educational
Number analyzed (Participants) | 20 | 21
units on a scale | -0.83 [-1.58 to -0.09] | -0.45 [-1.23 to 0.33]
Statistical Analysis 1: Comparison: Behavioral vs Educational; Test type: Superiority or Other; p = 0.47, Linear mixed model; Median Difference (Final Values) = -0.39, 95% CI 2-sided [-1.47 to 0.69]

2. Secondary Outcome: The Interference Subscale of the Multidimensional Pain Inventory (MPI)
Description: Secondary outcome is the estimated mean change in pain interference from baseline to 12 weeks post-baseline comparing CBT to Education.
  Pain Interference at the time of assessment; 0 = no interference to 6 = extreme interference. The higher the average number calculated for the subscale, the higher the perceived interference pain has on vocational, social/recreational, and family/martital functioning.
Time Frame: baseline to 12 weeks post-baseline [post-treatment]
Population: Not everyone that has baseline data completed 12-week post treatment data; making the number of participants analyzed different than reported for baseline data only.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Behavioral | Educational
Number analyzed (Participants) | 20 | 21
units on a scale | -0.03 [-0.58 to 0.52] | 0.31 [-0.28 to 0.91]
Statistical Analysis 1: Comparison: Behavioral vs Educational; baseline to 36 weeks post-baseline; Test type: Superiority or Other; p = 0.40, linear mixed model; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.15 to 0.47]

3. Secondary Outcome: Beck Depression Inventory (BDI)
Description: Estimated mean change in depressive symptoms from baseline to 12 weeks post-baseline combaring CBT and ED.
  0 (do not endorse) to 3 (highly endorse). no/minimal depressive symptoms =<10; mild-moderate depressive symptoms = 10-18; moderate-severe depressive symptoms = 19-29 severe depressive symptoms = 30-63. The higher the score, the more depressive symptoms endorsed.
Time Frame: baseline to 12 weeks post-baseline [post-treatment]
Population: Not everyone that has baseline data completed 12-week post treatment; making the number of participants analyzed differant than reported for baseline data only.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Behavioral | Educational
Number analyzed (Participants) | 20 | 21
units on a scale | -0.35 [-3.56 to 2.86] | 2 [-1.38 to 5.38]
Statistical Analysis 1: Comparison: Behavioral vs Educational; baseline to 12 weeks post-baseline; Test type: Superiority or Other; p = 0.31, Linear mixed model; Mean Difference (Final Values) = -2.35, 95% CI 2-sided [-7.02 to 2.32]

4. Primary Outcome: Numeric Rating Scale (NRS) Pain Intensity
Description: Primary outcome is the estimated mean change in pain intensity ratings from baseline to 36 weeks post-baseline comparing CBT and Educational arms
  Average pain intensity rating over the last 7 days; 0 (no pain at all) to 10 (worst pain imaginable); the higher the number, the greater percieved pain intensity.
Time Frame: baseline to 36 weeks post-baseline [follow-up]
Population: Not everyone that has baseline data completed 36-week follow up treatment data; making the number of participants analyzed different than reported for baseline data only.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Behavioral | Educational
Number analyzed (Participants) | 17 | 14
units on a scale | -0.87 [-1.58 to -0.17] | -0.89 [-1.65 to -0.12]
Statistical Analysis 1: Comparison: Behavioral vs Educational; baseline to 12 weeks comparison; Test type: Superiority or Other; p = 0.98, linear mixed model; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-1.03 to 1.06]

5. Secondary Outcome: The Interference Subscale of the Multidimensional Pain Inventory (MPI)
Description: Secondary outcome is the estimated mean change in pain interference from baseline to 36 weeks post-baseline comparing CBT to Education.
  Pain Interference at the time of assessment; 0 = no interference to 6 = extreme interference. The higher the average number calculated for the subscale, the higher the perceived interference pain has on vocational, social/recreational, and family/martital functioning.
Time Frame: baseline to 36 weeks post-baseline [follow-up]
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Behavioral | Educational
Number analyzed (Participants) | 17 | 14
units on a scale | 0.06 [-0.48 to 0.61] | 0.99 [0.35 to 1.62]
Statistical Analysis 1: Comparison: Behavioral vs Educational; baseline to 36 weeks post-baseline; Test type: Superiority or Other; p = 0.03, linear mixed model; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-1.76 to -0.07]

6. Secondary Outcome: Beck Depression Inventory (BDI)
Description: Estimated mean change in depressive symptoms from baseline to 36 weeks post-baseline comparing CBT to Education.
  0 (do not endorse) to 3 (highly endorse). no/minimal depressive symptoms =<10; mild-moderate depressive symptoms = 10-18; moderate-severe depressive symptoms = 19-29 severe depressive symptoms = 30-63. The higher the score, the more depressive symptoms endorsed
Time Frame: baseline to 36 weeks post-baseline [follow-up]
Population: Not everyone that has baseline data completed 36 week post treatment data; making the number of participants analyzed different than reported for baseline data only.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Behavioral | Educational
Number analyzed (Participants) | 17 | 14
units on a scale | .077 [-3.06 to 4.6] | 4.92 [0.7 to 9.15]
Statistical Analysis 1: Comparison: Behavioral vs Educational; baseline to 36 weeks post-baseline; Test type: Superiority or Other; p = 0.15, linear mixed model; Mean Difference (Final Values) = -4.16, 95% CI 2-sided [-9.86 to 1.55]

ADVERSE EVENTS:
Time Frame: AEs were collected weekly during the 10 week treatment program and again at 36 weeks during follow up.
Description: Occurances of AEs were asking at weekly treatment sessions and confirmed in the electronic medical record for the previous week of the session. During 36 week follow up, the electronic medical record was reviewed from the last treatment session to the current date of the assessment.
Arm/Group | Behavioral | Educational
Serious Adverse Events (participants affected / at risk) | 2/23 | 4/24
Other Adverse Events (participants affected / at risk) | 9/23 | 5/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral (N=23) | Educational (N=24)
Hyperglycemia (General disorders) | 1 (1) | 1 (1) — admission due to hyperglycemia Expected SAE for population
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Admission due to vehicular accident Unanticipated and unrelated SAE
Diabetic feet complications (Infections and infestations) | 0 (0) | 1 (2) — Admission due to diabetic feet complications Anticipated SAE for population
Thymectomy (Immune system disorders) | 0 (0) | 1 (1) — Unanticipated and unrelated SAE
Heart related issues (Cardiac disorders) | 1 (1) | 2 (2) — Chest pain, dyspnea Unanticipated and unrelated SAE
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral (N=23) | Educational (N=24)
Biopsy (Investigations) | 2 (2) | 1 (1) — biopsy of various systems (i.e. bladder, skin) - Unanticipated and unrelated AE
Infection (Infections and infestations) | 2 (2) | 1 (1) — Various infections (cellulitis, nausea, vomiting, flu-like symptoms - unanticipate and unrelated AE
Surgery or Procedure (Surgical and medical procedures) | 1 (1) | 1 (1) — Various surgeries or procedures (i.e. colonoscopy, submaxillary gland surgery) - Unanticipated and unrelated AE
ER due to pain (General disorders) | 4 (6) | 0 (0) — Mostly musculoskeletal (neck or leg pain) but also neurological (miagraine) - Unanticipated and unrelated AE
Hypoglycemia (General disorders) | 2 (2) | 0 (0) — non-admission, mild hypoglycemia - anticipated AE
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) — diagnosis of hepatitis C - Unanticipated and unrelated AE
Suicidal Ideation (SI) (Psychiatric disorders) | 0 (0) | 1 (1) — Endorses mild SI but after assessment from clinical psychologist, not deemed to be at risk - Unanticipated and unrelated AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No